CLINICAL TRIAL: NCT04544592
Title: Phase I/II Dose Escalation and Preliminary Efficacy of CD19 Directed CAR-T Cells Generated Using the Miltenyi CliniMACs Prodigy System (UCD19 CAR-T) in Pediatric Patients With Relapsed and/or Refractory B-Cell Acute Lymphoblastic Leukemia (B-ALL) and B-Cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: UCD19 CarT in Treatment of Pediatric B-ALL and B-NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-2424.cc; NCI-2020-08490 (Other: CTRP)
Record Dates: First submitted 2019-05-29; First posted 2020-09-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: Dose Escalation (Experimental): First 4-18 subjects enrolled. Treated with escalating doses of therapy until the recommended phase 2 dose (RP2D) is determined.
  Interventions: Drug: CD19CAR-CD3Zeta-4-1BB-Expressing Autologous T-Lymphocyte Cells
- Phase II: Dose Expansion (Experimental): Up to 18 additional subjects will be treated at the recommended Phase 2 dose (RP2D) to allow for 12 total subjects to be treated in each cohort, including those treated within the phase 1 portion.
  Interventions: Drug: CD19CAR-CD3Zeta-4-1BB-Expressing Autologous T-Lymphocyte Cells

INTERVENTIONS:
Drug: CD19CAR-CD3Zeta-4-1BB-Expressing Autologous T-Lymphocyte Cells — The CD19 CAR used in this study consists of three main components: the variable regions of the anti-CD19 monoclonal antibody FMC63 71, linked to the TNFRSF-19-derived transmembrane domain, the 4-1BB costimulatory molecule, and the signaling domain of the CD3-zeta molecule. The DNA encoding this receptor was cloned into a lentiviral vector (LV) backbone.

SUMMARY:
This phase I/II trial will investigate a new CD19 directed CAR-T therapy manufactured locally with the goals to expedite infusion to wider patient inclusion that includes those who were previously excluded, such as pediatric patients with B-cell NHL and patients in primary relapse.

DETAILED DESCRIPTION:
Pediatric patients with refractory or multiply relapsed leukemia and lymphoma do poorly with traditional chemotherapy and have overall survival rates below 20%-50% depending on a variety of disease and patient related characteristics. Approximately 10-20% of pediatric patients with pre B-ALL will relapse (1) and relapsed pre B-ALL is a leading cause of cancer death in children (2). Site of relapse and timing of first relapse from initial therapy are important factors that impact the survival rates after first relapse (3). The 5-year survival for pre B-ALL pediatric patients with early relapse is 25-50% (2). Pediatric patients who experience a late relapse have excellent survival rates with chemotherapy alone, however if they have MRD positivity after reinduction, this drops their survival rates down to 50-60% (4). The FDA approval of CD19-directed CAR-T cell therapy has increased treatment options for patients with refractory disease or those in second relapse. However, many patients, including those in first relapse do not fit the current criteria to receive this treatment. As well, regardless of the number of prior relapses, some patients in second relapse cannot tolerate the extended delay and ongoing therapy that is necessary for the commercial manufacturing of these cells at the commercial level.

This phase I/II trial will investigate a new CD19-directed CAR-T therapy manufactured locally with the goal of expediting the infusion to patients who were previously excluded, such as pediatric patients with relapsed B-cell NHL and patients in their initial (or greater) leukemic relapse. We hypothesize that CD19-directed CAR-T cells manufactured using the Miltenyi CliniMACs Prodigy System (UCD19 CAR-T) will be safe, well-tolerated, and show preliminary efficacy in pediatric patients with relapsed and/or refractory B-ALL or B-NHL. No controls will be used beyond historical comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Meets clinical criteria for leukapheresis or has a leukapheresis product previously collected and stored per recommended guidelines.
2. Provision of signed and dated consent form from parent or guardian (patients <18), the patient themselves (>18), or legally authorized representative (patient >18 who lack decision-making capacity); Pediatric patients will be included in age-appropriate discussions and assent will be obtained for those > 7 years of age, when appropriate, according to institutional standards.
3. Willingness to participate in long term follow up study.
4. Stated willingness to comply with all study procedures and be available for the duration of the study.
5. Males OR non-pregnant, non-breastfeeding females.

   o Patients of child-bearing potential or capable of fathering a child must agree to use highly effective contraception from the time of initial CAR T cell administration though 12 months following the final administration of investigational product.
6. Aged 31 days to 30 years (inclusive) at time of consent and enrollment.
7. Acute Lymphoblastic Leukemia (ALL) OR Non-Hodgkin Lymphoma (NHL) of B-cell origin that:

   o Has confirmed expression of CD19 by flow cytometry, immunohistochemistry (IHC), or both.

   Cohort One Criteria:
   * Meets any one of the following conditions:

     * Relapsed two or more times
     * Relapsed at any time after allogeneic BMT
     * Refractory to standard therapy as determined by the treating physician
     * Meets criteria for BMT but is ineligible as determined by the treating physician
     * Patient and/or parents declining BMT options and would prefer CAR-T Therapy.
   * Non-Hodgkin Lymphoma includes all of the following:

     * Diffuse large B-cell lymphoma (DLBCL)
     * Burkitt Lymphoma
     * Intermediate lymphoma between Burkitt and DLBCL
     * Primary Mediastinal B-cell Lymphoma (PMBL)
     * Follicular lymphoma
     * High grade B cell lymphoma
     * Transformed lymphoma

   Cohort Two Criteria:
   * B-ALL in first relapse with any one of the following conditions:

     * High-risk genomic alterations at initial diagnosis such as KMT2A gene rearrangement, t(17;19), hypodiploidy, Ph-like mutations, BCR-ABL1 fusion (Ph+ ALL), iAMP21, and TP53 inactivating mutation/deletion.
     * Isolated CNS relapse such that cranial radiation would be indicated as a component of standard salvage therapy.
     * Down syndrome.
     * Minimal residual disease (MRD) positivity of > 0.01% by FACS or > 0 clonal sequences by NGS in bone marrow post re-induction chemotherapy.
     * Age 18 years or older. OR
   * Newly diagnosed with persistent MRD ≥ 0.01% by flow cytometry in bone marrow at end of consolidation.
8. Performance score (Lansky or Karnofsky) of 50% or better;
9. Unable to or declined to receive commercially available CD19 CAR-T Therapy.

Exclusion Criteria:

1. Evidence of rapidly progressive disease without adequate salvage/bridging regimens as determined by the investigator.
2. Active Graft-versus-Host Disease (GvHD).
3. Active, uncontrolled, life-threatening infection that at the determination of the treating physician would preclude safe leukapheresis or tolerance of LD chemotherapy, cell infusion, or cytokine release syndrome.
4. Evidence of severe organ dysfunction as defined by:

   * Myocardial dysfunction: Ejection fraction ≤ 40% or shortening fraction ≤ 28%, evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO), and clinically significant electrocardiogram (ECG) findings.
   * Baseline oxygen saturation of ≤ 90% on room air
   * Transaminases > 10x upper limit of normal (ULN) or bilirubin >2x the ULN, unless thought to be related to primary disease
   * Estimated Cr clearance <60 mL/min/1.73 m2 (if nuclear medicine GFR or other more specific testing exceeds this level than it can supersede the estimated clearance)
5. Post-pubertal females that are pregnant, planning to become pregnant, or unwilling to use birth control (includes abstinence) for the study duration.
6. Known HIV infection, or active Hepatitis B or active Hepatitis C infection.
7. Prior gene therapy, including prior CAR-T cell.

Ages: 31 Days to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and tolerability of UCD19 CAR-T infusion in pediatric patients with B-ALL or B-NHL | Post UCD19 infusion to Day 28
  DLTs of UCD19 CAR-T will be assessed at each of the dose levels in a standard 3+3 dose-escalation design with a determination of recommended Phase 2 dose (RP2D).
Determine the preliminary efficacy of UCD19 CAR-T cells in pediatric patients with B-ALL or B-NHL | Day 28 (for B-ALL) and Day 90 (for B-NHL) post UCD19 infusion
  Following determination of UCD19 CAR-T RP2D, there will be a cohort expansion to determine preliminary efficacy and biological activity by assessment of CR status.

SECONDARY OUTCOMES:
Determine the preliminary efficacy of UCD19 CAR-T cells in pediatric patients with B-ALL during the expansion phase | Day 60
  Rate of patients who have morphologic remission post infusion for B-ALL as assessed by bone marrow morphology.
Determine the preliminary efficacy of UCD19 CAR-T cells in pediatric patients with B-ALL during the expansion phase | Day 90
  Rate of patients with radiographic remission post infusion for B-NHL
Determine the preliminary efficacy of UCD19 CAR-T cells in pediatric patients with B-ALL during the expansion phase | Months 1, 2, 3, 6, and 12
  Rate of efficacy as assessed by bone marrow minimal residual disease assessment by flow cytometric analysis and next generation sequencing for B-ALL patients
Determine the preliminary efficacy of UCD19 CAR-T cells in pediatric patients with B-ALL during the expansion phase | Months 1, 2, 3, 6, and 12
  Median duration of remission as assessed by bone marrow minimal residual disease assessment by flow cytometric analysis and next generation sequencing for B-ALL patients
Determine the preliminary efficacy of UCD19 CAR-T infusion in pediatric patients after first relapse with B-ALL during the expansion phase | At Months 6 and 12
  Rate of event free survival (EFS) post UCD19 CAR-T cell infusion for B-ALL patients in first relapse.
Determine the preliminary efficacy of UCD19 CAR-T infusion in pediatric patients after first relapse with B-ALL during the expansion phase | At Months 1, 2 , 3, 6 and 12-months
  Median duration of B-cell aplasia will be assessed by flow cytometry post UCD19 CAR-T cell infusion.
Determine the preliminary efficacy of UCD19 CAR-T infusion in pediatric patients after first relapse with B-ALL during the expansion phase | Up to 12 months post infusion
  Incidence of patients who require stem cell transplantation (SCT) within 12-months post UCD19 CAR-T cell infusion.
Determine the preliminary efficacy of UCD19 CAR-T infusion in pediatric patients after first relapse with B-ALL during the expansion phase | Up to 12 months post infusion
  Incidence of patients who require cranial radiation within 12-months post UCD19 CAR-T cell infusion.
Determine the preliminary efficacy of UCD19 CAR-T infusion in pediatric patients after first relapse with B-ALL during the expansion phase | Up to 12 months post infusion
  Incidence of clinically significant infections (defined as those that require treatment) will be collected over the first year of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Fabrizio, MD, MS, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No